CLINICAL TRIAL: NCT00369057
Title: Intra Ocular Pressure During Robotic Prostatectomy
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 0510008190
Record Dates: First submitted 2006-08-25; First posted 2006-08-29 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Visual Acuity; Visual Disturbance; Intraocular Pressure
Keywords: Intraocular pressure; Prostatectomy; Robotic; Glaucoma; Carbon dioxide
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Our goal is to study the relationship between intraocular pressure during robotic prostatectomy surgery and visual deficiencies/vision loss after surgery. We believe the risk of vision loss from this surgery to be due to positioning during the operation, as well as abdominal carbon dioxide insufflation. As robotic procedures are gaining in popularity, we should determine whether they are subjecting this patient population, and perhaps more likely the patient with a preoperative diagnosis of glaucoma, to an increased likelihood of postoperative visual disturbance.If our hypothesis that intraocular pressure is increased in these patients is confirmed, future studies will assess therapeutic modalities to maintain the IOP near baseline.

DETAILED DESCRIPTION:
The frequency of post-operative permanent vision loss has been recently estimated to be 1:61,0001,2 , although the majority of these cases involve surgical trauma to the eye or brain. Prolonged vision loss not attributable to direct trauma has been estimated to occur with a frequency of approximately 1:125,0003 and has been given a broad classification termed ischemic optic neuropathy. This rare but catastrophic outcome has most commonly been associated with operations performed under circumstances in which there may be increased intraocular pressure (IOP), either due to positioning4 or due to insufflation of the abdomen with carbon dioxide (laparoscopy).5

There are two factors predisposing the robotic prostatectomy patient to an increase in IOP: step head-down (Trendelenburg) position and abdominal carbon dioxide (CO2) insufflation. The Trendelenburg position will increase central venous pressure within the thorax, which may reduce the drainage of blood flow from the head, thus increasing IOP. The CO2 insufflation may increase IOP via two mechanisms. First, by increasing intra-abdominal pressure there is a further increase in intrathoracic pressure. Secondly, insufflation the CO2 may increase the carbon dioxide content of the blood, to which the brain reacts by vasodilating and increasing blood volume. Thus while flow into the eye is increased, flow out of the eye is decreased leading to an increase in pressure inside the eye which eventually may reduce the inflow enough to cause retinal or optic nerve ischemia.

Because the pressure within the eye is an important factor in determining the blood flow to the eye, prevention of a dramatic increase in IOP may make patients less vulnerable to peri-operative ischemic optic neuropathy and vision loss. Because permanent vision loss is such a rare event after surgery, this study will measure more subtle (and most likely, temporary) vision changes (subjective blurriness, visual field deficits, decreased acuity), which occur more frequently and are thus a more easily measured outcome.6

As robotic procedures are gaining in popularity, we should determine whether they are subjecting this patient population, and perhaps more likely the patient with a preoperative diagnosis of glaucoma, to an increased likelihood of postoperative visual disturbance.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 18 or older
* Scheduled for Robotic Prostatectomy Surgery
* ASA Classification of I, II, or III
* Good comprehension of written and spoken english.

Exclusion Criteria:

* Allergy to Tetracaine or related anesthetics
* Glaucoma
* Asthma
* History of heart electrical problems

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult males aged 18 or older, undergoing robotic prostatectomy at NewYork Presbyterian Hospital with no pre-existing eye conditions.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2006-02; Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Fogarty-Mack, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States